CLINICAL TRIAL: NCT02989389
Title: Single-Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3323795 in Healthy Subjects
Brief Title: A Study of LY3323795 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16610; I9F-MC-SCAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Results first posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LY3323795 (Part A) (Experimental): Participants received escalating doses of 0.3 mg (milligrams), 1 mg, 3 mg, 10 mg, 30 mg and 100 mg of LY3323795 orally.
  Interventions: Drug: LY3323795
- Placebo (Part A) (Placebo Comparator): Participants received placebo identical to LY3323795 orally.
  Interventions: Drug: Placebo
- LY3323795 (Part B) (Experimental): Participants received 6 mg, 20 mg and 80 mg of LY3323795 orally.
  Interventions: Drug: LY3323795
- Placebo (Part B) (Placebo Comparator): Participants received placebo identical to LY3323795 orally.
  Interventions: Drug: Placebo
- LY3323795 (Part C) (Experimental): Part C was not initiated due to a Lilly internal strategy decision.
  Interventions: Drug: LY3323795
- LY3323795 + Itraconazole (Part C) (Experimental): Part C was not initiated due to a Lilly internal strategy decision.
  Interventions: Drug: LY3323795; Drug: Itraconazole

INTERVENTIONS:
Drug: LY3323795 — Administered orally
  Arms: LY3323795 (Part A); LY3323795 (Part B); LY3323795 (Part C); LY3323795 + Itraconazole (Part C)
Drug: Itraconazole — Administered orally
  Arms: LY3323795 + Itraconazole (Part C)
Drug: Placebo — Administered orally
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to investigate the safety of LY3323795 and the effects it has on the body. The study drug or placebo (sugar pill) will be given by mouth to healthy participants. The study has three parts. Each participant may only enroll in one part. The study will last 14 to 43 days, depending on the part. Screening must be completed prior to study start.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of non-childbearing potential at time of screening
* Have a body mass index (BMI) between 18.0 kilograms per square meter (kg/m²) and 32.0 kg/m², inclusive

Exclusion Criteria:

* Have participated, within the last 30 days, in a clinical trial involving an investigational product.
* Have a QT corrected for heart rate (QTc) (using Bazett's formula) interval value of greater than 450 millisecond (msec) (males) or greater than 470 msec (females)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A was a dose-escalation 3-period crossover with 2 alternating cohorts (Cohorts 1 and 2). There was 14 days of washout time between each dose. Part B was a single-dose, 3-cohort (Cohorts 3, 4 and 5) study.
Groups:
- Part A-Cohort 1 (Sequence 1): Participants received 0.3 milligrams (mg), 3 mg, 30 mg LY3323795 and Placebo. Period 1: Placebo, Period 2: 3 mg LY3323795, Period 3: 30 mg LY3323795
- Part A-Cohort 1 (Sequence 2): Participants received 0.3 mg, 3 mg, 30 mg LY3323795 and Placebo. Period 1: 0.3 mg LY3323795, Period 2: Placebo, Period 3: 30 mg LY3323795
- Part A-Cohort 1 (Sequence 3): Participants received 0.3 mg, 3 mg, 30 mg LY3323795 and Placebo. Period 1: 0.3 mg LY3323795, Period 2: 3 mg LY3323795, Period 3: Placebo
- Part A-Cohort 2 (Sequence 1): Participants received 1 mg, 10 mg, 100 mg of LY3323795 and Placebo. Period 1: 1 mg LY3323795, Period 2: 10 mg LY3323795, Period 3: Placebo
- Part A-Cohort 2 (Sequence 2): Participants received 1 mg, 10 mg, 100 mg of LY3323795 and Placebo. Period 1: Placebo, Period 2: 10 mg LY3323795, Period 3: 100 mg LY3323795
- Part A-Cohort 2 (Sequence 3): Participants received 1 mg, 10 mg, 100 mg of LY3323795 and Placebo. Period 1: 1 mg LY3323795, Period 2: Placebo, Period 3: 100 mg LY3323795
- Part B, 6 mg LY3323795: Participants received 6 mg of LY3323795 orally.
- Part B, 20 mg LY3323795: Participants received 20 mg of LY3323795 orally.
- Part B, 80 mg LY3323795: Participants received 80 mg of LY3323795 orally.
- Part B, Placebo: Participants received placebo identical to LY3323795 orally.
Period: Period 1
Arm/Group | Part A-Cohort 1 (Sequence 1) | Part A-Cohort 1 (Sequence 2) | Part A-Cohort 1 (Sequence 3) | Part A-Cohort 2 (Sequence 1) | Part A-Cohort 2 (Sequence 2) | Part A-Cohort 2 (Sequence 3) | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Part B, Placebo
Started | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 6
Received at Least 1 Dose of Study Drug | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 6
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 5 | 5 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Part A-Cohort 1 (Sequence 1) | Part A-Cohort 1 (Sequence 2) | Part A-Cohort 1 (Sequence 3) | Part A-Cohort 2 (Sequence 1) | Part A-Cohort 2 (Sequence 2) | Part A-Cohort 2 (Sequence 3) | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Part B, Placebo
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 (Part B was planned as a single period study.) | 0 (Part B was planned as a single period study.) | 0 (Part B was planned as a single period study.) | 0 (Part B was planned as a single period study.)
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A-Cohort 1 (Sequence 1) | Part A-Cohort 1 (Sequence 2) | Part A-Cohort 1 (Sequence 3) | Part A-Cohort 2 (Sequence 1) | Part A-Cohort 2 (Sequence 2) | Part A-Cohort 2 (Sequence 3) | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Part B, Placebo
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A-Cohort 1 (Sequence 1) | Part A-Cohort 1 (Sequence 2) | Part A-Cohort 1 (Sequence 3) | Part A-Cohort 2 (Sequence 1) | Part A-Cohort 2 (Sequence 2) | Part A-Cohort 2 (Sequence 3) | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Part B, Placebo | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 6 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 4 | 6 | 6 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 2 | 1 | 2 | 11
  Male | 3 | 4 | 2 | 3 | 1 | 3 | 3 | 3 | 5 | 4 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 9
  Not Hispanic or Latino | 1 | 3 | 2 | 2 | 2 | 1 | 5 | 5 | 6 | 5 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 10
  White | 3 | 1 | 2 | 2 | 2 | 2 | 5 | 3 | 3 | 3 | 26
  More than one race | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 6 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Data presented are the number of participants who experienced 1 or more SAEs considered by the investigator to be related to study drug administration is reported. SAEs were classified using the Medical Dictionary for Regulatory Activities (MedDRA) 19.1. A summary of non-serious adverse events and all serious adverse events, regardless of causality is located in the Reported Adverse Events section.
Time Frame: Baseline to Study Completion (up to Day 43)
Population: All randomized participants who received study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A, Cohort 1, Placebo; Part A, Cohort 2, Placebo; Part B, Placebo: Participants received placebo identical to LY3323795 orally.
- Part A, Cohort 1, 0.3 mg LY3323795: Participants received 0.3 mg of LY3323795 orally.
- Part A, Cohort 1, 3 mg LY3323795: Participants received 3 mg of LY3323795 orally.
- Part A, Cohort 1, 30 mg LY3323795: Participants received 30 mg of LY3323795 orally.
- Part A, Cohort 2, 1 mg LY3323795: Participants received 1 mg of LY3323795 orally.
- Part A, Cohort 2, 10 mg LY3323795: Participants received 10 mg of LY3323795 orally.
- Part A, Cohort 2, 100 mg LY3323795: Participants received 100 mg of LY3323795 orally.
Arm/Group | Part A, Cohort 1, Placebo | Part A, Cohort 1, 0.3 mg LY3323795 | Part A, Cohort 1, 3 mg LY3323795 | Part A, Cohort 1, 30 mg LY3323795 | Part A, Cohort 2, Placebo | Part A, Cohort 2, 1 mg LY3323795 | Part A, Cohort 2, 10 mg LY3323795 | Part A, Cohort 2, 100 mg LY3323795 | Part B, Placebo | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3323795 in Plasma
Description: Pharmacokinetics (PK): Maximum observed drug concentration (Cmax) of LY3323795 in plasma.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72,96,120,144 hours, post dose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A, Cohort 1, 0.3 mg LY3323795 | Part A, Cohort 2, 1 mg LY3323795 | Part A, Cohort 1, 3 mg LY3323795 | Part A, Cohort 2, 10 mg LY3323795 | Part A, Cohort 1, 30 mg LY3323795 | Part A, Cohort 2, 100 mg LY3323795 | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6
nanogram per milliliter (ng/mL) | 0.503 (32) | 1.77 (29) | 4.79 (24) | 15.7 (25) | 34.6 (35) | 89.1 (44) | 10.4 (45) | 27.2 (26) | 88.1 (34)

3. Secondary Outcome: Part B Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3323795 in Cerebrospinal Fluid (CSF)
Description: Part B Pharmacokinetics (PK): Maximum observed drug concentration (Cmax) of LY3323795 in cerebrospinal fluid (CSF).
Time Frame: -4, -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36 hours, post dose
Population: All randomized participants from Part B group, who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795
Number analyzed (Participants) | 6 | 5 | 6
nanogram per milliliter (ng/mL) | 0.293 (31) | 0.788 (11) | 2.86 (34)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time Zero to Tlast (AUC[0-tlast]) of LY3323795 in Plasma
Description: Pharmacokinetics (PK): Area under the concentration time curve from time zero to tlast (AUC[0-tlast]) of LY3323795 in plasma.
Time Frame: 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72,96,120,144 hours, post dose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- Part A, Cohort 1, 30 mg LY3323795: Participants received 10 mg of LY3323795 orally.
Arm/Group | Part A, Cohort 1, 0.3 mg LY3323795 | Part A, Cohort 2, 1 mg LY3323795 | Part A, Cohort 1, 3 mg LY3323795 | Part A, Cohort 2, 10 mg LY3323795 | Part A, Cohort 1, 30 mg LY3323795 | Part A, Cohort 2, 100 mg LY3323795 | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 7 | 6
nanogram*hour per milliliter (ng*h/mL) | 5.67 (69) | 25.2 (28) | 73.4 (31) | 274 (14) | 663 (35) | 2370 (29) | 156 (17) | 441 (24) | 1950 (49)

5. Secondary Outcome: Part B Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time Zero to Tlast (AUC[0-tlast]) of LY3323795 in Cerebrospinal Fluid (CSF)
Description: Part B Pharmacokinetics (PK): Area under the concentration time curve from time zero to tlast (AUC[0-tlast]) of LY3323795 in cerebrospinal fluid (CSF).
Time Frame: -4, -2, 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36 hours, post dose
Population: All randomized participants from Part B group, who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795
Number analyzed (Participants) | 6 | 5 | 6
ng*h/mL | 5.46 (24) | 13.7 (16) | 55.1 (48)

6. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Plasma Amyloid Beta (Aβ)₁-₄₀ and Aβ₁-₄₂
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein, plasma concentrations of Aβ1-40 and Aβ1-42 were determined using validated immunoassay methods.
Time Frame: Baseline through 144 hours
Population: All randomized participants who received at least 1 dose of study drug and have baseline and at least one post-baseline plasma Aβ1-40 or Aβ1-42 data.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/mL)
Groups:
- Placebo: Participants received placebo identical to LY3323795 orally.
Arm/Group | Part A, Cohort 1, 0.3 mg LY3323795 | Part A, Cohort 2, 1 mg LY3323795 | Part A, Cohort 1, 3 mg LY3323795 | Part A, Cohort 2, 10 mg LY3323795 | Part A, Cohort 1, 30 mg LY3323795 | Part A, Cohort 2, 100 mg LY3323795 | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 24
Picogram per milliliter (pg/mL)
  Aβ1-40 | -39 (8) | -52 (6) | -71 (7) | -76 (4) | -76 (18) | -89 (2) | -79 (7) | -81 (5) | -89 (1) | -23 (11)
  Aβ1-42 | -22 (7) | -33 (6) | -49 (5) | -60 (5) | -63 (8) | -75 (3) | -54 (11) | -58 (6) | -64 (9) | -12 (6)

7. Secondary Outcome: Part B Pharmacodynamics (PD): Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid Beta (Aβ)₁-₄₀ and Aβ₁-₄₂
Description: Amyloid beta is a peptide fragment of the amyloid precursor protein, CSF concentrations of Aβ1-40, Aβ1-42 were determined using validated immunoassay methods.
Time Frame: Baseline through 36 hours
Population: All randomized participants from Part B group, who received at least 1 dose of study drug and have baseline and at least one post-baseline CSF Aβ1-40 or Aβ1-42 data.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/mL)
Arm/Group | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Placebo
Number analyzed (Participants) | 6 | 5 | 4 | 6
Picogram per milliliter (pg/mL)
  Aβ 1-40 | -51 (21) | -69 (6) | -88 (4) | -12 (11)
  Aβ 1-42 | -37 (23) | -71 (10) | -81 (7) | -17 (23)
Statistical Analysis 1: Comparison: Part B, 6 mg LY3323795 vs Placebo; Aβ 1-40; Test type: Superiority; p = 0.215, Mixed Models Analysis; Mean Difference (Final Values) = -11.57, 90% CI 2-sided [-29.52 to 10.96]
Statistical Analysis 2: Comparison: Part B, 20 mg LY3323795 vs Placebo; Aβ 1-40; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -60.53, 90% CI 2-sided [-69.79 to -48.43]
Statistical Analysis 3: Comparison: Part B, 80 mg LY3323795 vs Placebo; Aβ 1-40; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -87.07, 90% CI 2-sided [-90.21 to -82.92]
Statistical Analysis 4: Comparison: Part B, 6 mg LY3323795 vs Placebo; Aβ 1-42; Test type: Superiority; p = 0.015, Mixed Models Analysis; Mean Difference (Final Values) = -19.60, 90% CI 2-sided [-33.69 to -2.51]
Statistical Analysis 5: Comparison: Part B, 20 mg LY3323795 vs Placebo; Aβ 1-42; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -65.41, 90% CI 2-sided [-72.23 to -56.92]
Statistical Analysis 6: Comparison: Part B, 80 mg LY3323795 vs Placebo; Aβ 1-42; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -84.56, 90% CI 2-sided [-88.97 to -78.38]

ADVERSE EVENTS:
Time Frame: Up to 43 days
Description: All enrolled participants who received study drug.
Arm/Group | Part A, Cohort 1, Placebo | Part A, Cohort 1, 0.3 mg LY3323795 | Part A, Cohort 1, 3 mg LY3323795 | Part A, Cohort 1, 30 mg LY3323795 | Part A, Cohort 2, Placebo | Part A, Cohort 2, 1 mg LY3323795 | Part A, Cohort 2, 10 mg LY3323795 | Part A, Cohort 2, 100 mg LY3323795 | Part B, 6 mg LY3323795 | Part B, 20 mg LY3323795 | Part B, 80 mg LY3323795 | Part B, Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 2/6 | 0/6 | 0/6 | 1/9 | 1/6 | 0/6 | 2/6 | 5/6 | 3/5 | 6/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, Cohort 1, Placebo (N=9) | Part A, Cohort 1, 0.3 mg LY3323795 (N=6) | Part A, Cohort 1, 3 mg LY3323795 (N=6) | Part A, Cohort 1, 30 mg LY3323795 (N=6) | Part A, Cohort 2, Placebo (N=9) | Part A, Cohort 2, 1 mg LY3323795 (N=6) | Part A, Cohort 2, 10 mg LY3323795 (N=6) | Part A, Cohort 2, 100 mg LY3323795 (N=6) | Part B, 6 mg LY3323795 (N=6) | Part B, 20 mg LY3323795 (N=5) | Part B, 80 mg LY3323795 (N=6) | Part B, Placebo (N=6)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Part C (an itraconazole interaction study) was not initiated due to a Lilly internal strategy decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT02989389/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02989389/SAP_001.pdf